CLINICAL TRIAL: NCT00671411
Title: Evaluation of Renal Masses Using Ultrasound Intravenous Microbubble Contrast
Brief Title: Evaluating Renal Masses Using Ultrasound Intravenous Microbubble Contrast
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 07-165
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Renal Cancer; Kidney Cancer
Keywords: Ultrasound; 07-165
MeSH Terms: conditions — Kidney Neoplasms | interventions — High-Energy Shock Waves; Congresses as Topic; Amino Acid Motifs

ARMS (1):
- 1 (Experimental): Patients entering into this protocol will also have a preoperative renal contrast enhanced US for this research study. Renal mass US contrast enhancement results will be compared with surgical pathological findings to determine if contrast enhancement patterns of the renal masses correlate with benign and malignant histopathology, and/or malignant histologic subtype.
  Interventions: Drug: Ultrasound with intravenous microbubble contrast injection

INTERVENTIONS:
Drug: Ultrasound with intravenous microbubble contrast injection — Intravenous line will be inserted. After the ultrasound microbubble contrast has been suspended into solution, contrast will be injected intrav via hand bolus with a total activated suspension of 0.2 mL (30 uL octaflouropropane),followed by 10 mL saline flush, with option to rebolus 4 addit time's for tot dose of 150 uL. Post contrast cine images of renal mass will be obtained on commercially available US units primarily using low mechanical index settings & Contrast Pulsed Sequence (CPS®) technique. Images will be acquired at predetermined intervals, for up to 8 min post contrast admin. Manufacturer's guidelines incl immediate post flush image capture, as well as post admin image capture at intervals as 1 min, 2 , 4 & 8 mins. Additional, temporary higher mechanical index imaging of kidney for the purpose of "flash" bubble destruction may be optionally triggered using manufacturer's preset settings & energy w/i FDA guidelines. This will only be performed while imaging the kidney.
  Other Names: Conventional and contrast enhanced US images will be saved to the hard drive; and /or digitally archived, without any unique identifiers, and reviewed at a; later date. Images will be reviewed by three radiologists who are blinded to; the clinical, pathologic, and non ultrasound imaging findings. Grayscale; characteristics, qualitative and quantitative enhancement characteristics will; be recorded.

SUMMARY:
The purpose of this study is to evaluate the blood flow in kidney masses by using ultrasound microbubble contrast material, and to see if results from ultrasound contrast studies can predict if a kidney mass is benign or malignant. Patterns of blood flow in the kidney mass will be examined to see if:

1. benign kidney masses can be distinguished from kidney cancers and
2. if slow growing, lower risk cancers have different blood flow compared to clear cell cancer which is the most common type of kidney cancer.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient who is planned or scheduled for surgical excision or biopsy of a solid or complex cystic renal mass would be eligible for the study
* Histology of the renal mass must be unknown at the time of enrollment
* Patients who have renal masses that are evident on conventional US imaging
* Patients will have a correlative abdominal CT and/or MRI

Exclusion Criteria:

* Patients with any history of cardiac shunts.
* Patients with history of pulmonary hypertension or unstable cardiopulmonary conditions, including patients on mechanical ventilation.
* Patients without peripheral IV access
* Pregnant patients and children
* Patients with any known contrast allergies, allergy to perflutren, or any components of Definity or microbubble contrast
* Patients who have renal masses that are not evident on conventional US imaging

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To determine the accuracy of contrast enhanced ultrasound of renal masses to predict benign vs. malignant histology | conclusion of study

SECONDARY OUTCOMES:
To determine if clear cell renal malignancies can be predicted, or differentiated, from other less aggressive malignant subtypes, based on analysis of the data. | conclusion of study
To determine if contrast enhanced ultrasound of renal masses provides added value in predicting benign vs. malignant histology, when compared to the current routine evaluation of CT or MRI, and standard grey scale and Doppler US | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Scott Gerst, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org